CLINICAL TRIAL: NCT03856606
Title: The Effects of Interrupting Prolonged Sitting With Intermittent Exercise on Postprandial Lipemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Edward F. Coyle, Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2017-11-0141
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Metabolic Syndrome X; Atherosclerosis; Insulin Resistance; Hyperinsulinism; Glucose Metabolism Disorders; Metabolic Disease; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Metabolic Syndrome; Atherosclerosis; Insulin Resistance; Hyperinsulinism; Glucose Metabolism Disorders; Metabolic Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged sitting without exercise (Experimental): Subjects will be asked to undergo prolonged sitting (~14 hours) of 1 day and will not be asked to perform interval exercise.
  Interventions: Behavioral: Prolonged sitting without exercise
- Prolonged sitting with interval exercise (Experimental): Subjects will be asked to undergo prolonged sitting (~14 hours) of 1 day and will be asked to perform interval exercise every hour on the hour.
  Interventions: Behavioral: Prolonged sitting with interval exercise

INTERVENTIONS:
Behavioral: Prolonged sitting without exercise — Subjects will have a 2-day control period during which step count and diet will be controlled for and recreated for the other trial. Following this 2-day period, they will undergo the prolonged sitting trial. Day 4 will consist of the lipid tolerance test to determine the ability of the body to clear triglycerides.
  Arms: Prolonged sitting without exercise
Behavioral: Prolonged sitting with interval exercise — Subjects will have a 2-day control period during which step count and diet will be controlled for and recreated for the other trial. Following this 2-day period, they will undergo a prolonged sit which with will be broken up every hour on the hour by a small bout of interval exercise. Day 4 will consist of the lipid tolerance test to determine the ability of the body to clear triglycerides.
  Arms: Prolonged sitting with interval exercise

SUMMARY:
The purpose of this study is to investigate the effect of interrupting prolong sedentary behavior with interval exercise on postprandial metabolism following a high fat glucose tolerance test.

DETAILED DESCRIPTION:
All subjects complete two trials in a randomized crossover design, with each trial occurring over 4 days with a minimum of seven days between trials. The first two days of each trial serve as a control period allowing for familiarization and the control of physical activity and calorie consumption prior to the intervention. Following each control period, subjects then perform one of the interventions on Day 3. The interventions consist of either eight-hours of prolonged sitting, or eight hours of sitting interrupted every hour by five sprints lasting 4 seconds each using the interval exercise. On day 4, all subjects will undergo a high fat glucose tolerance test to determine the body's ability to clear triglycerides from the blood as well as insulin/glucose response and substrate oxidation. Blood samples will be assayed for the previously mentioned substances and postprandial gas collection will be analyzed via indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* cardiovascular problems (e.g. pre-existing heart issues, coronary artery disease, hypertension, etc.)
* respiratory problems
* musculoskeletal problems that prevent prolonged sitting or exercise
* susceptibility to fainting
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-07-08 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
Plasma Triglycerides | 6-hours
  Areas under the curve for triglyceride concentration will be calculated for hourly samples from a 6-hour lipid tolerance test

SECONDARY OUTCOMES:
Plasma Insulin | 6-hours
  Areas under the curve for insulin concentration will be calculated for hourly samples from a 6-hour lipid tolerance test
Plasma Glucose | 6-hours
  Areas under the curve for glucose concentration will be calculated for hourly samples from a 6-hour lipid tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Coyle, Ph.D., Study Director — University of Texas at Austin
Locations (1):
- University of Texas at Austin Human Performance Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No